CLINICAL TRIAL: NCT01725763
Title: Non-contrast Enhanced Cardiac Magnetic Resonance Imaging in the Diagnosis and Classification of Pulmonary Hypertension
Acronym: CMR-PH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Ursula Reiter, Principal Investigator, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMR-12-PH
Record Dates: First submitted 2012-11-03; First posted 2012-11-14 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Hypertension; Elevated Mean Pulmonary Arterial Pressure; Normal Mean Pulmonary Arterial Pressure
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- suspected PH (Other): 60 minute Cardiac MRI
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI

SUMMARY:
Pulmonary hypertension (PH) is a life-threatening cardiovascular disease characterized by pathological elevation of mean pulmonary arterial pressure (mPAP) >/= 25 mmHg at rest. mPAP < 20 mmHg is defined as normal, values in the range between 21-24 mmHg are described as "borderline PH" diagnosed by right heart catheterization. Based on the etiology, PH is assigned to 5 groups (WHO, Data Point, 2008), whereas classification of disease is an important prognostic and therapy-deciding criterion.

Cardiac magnetic resonance tomography (CMR) provides a reliable technique to estimate elevated mean pulmonary arterial pressure from period of existence of a vortical motion of blood flow in the main pulmonary artery. Vortex can be visualized in 3-dimensional vector field, particle trace and streamline representations and can be analysed with respect to vortex related measures (geometry of center, vortex formation, vorticity, propagation dynamics …). Furthermore T1-mapping and non-contrast enhanced lung perfusion/ventilation scans represent promising techniques for PH characterization.

Aim of this explorative study is to 1. analyse PH-associated blood flow characteristics in the heart and the surrounding great vessels with respect to the 5 groups of PH, and 2. investigate the hemodynamic state of "borderline PH" compared to normal mPAP and manifest PH by non-contrast CMR.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected or known PH scheduled for routine right-heart catheterization,
* ability to give informed consent.

Exclusion Criteria:

* General MR exclusion criteria eg. patients with metal devices or other magnetic material in or on the subjects body which will be hazardous for MR investigation (e.g. heart pace-maker, brain aneurysm clip, nerve stimulators, electrodes, penile implants, coloured contact lenses, patch to deliver medications through the skin, any metal implants as rods, joints, plates, pins, screws, nails or clips, embolization coil, or any metal fragments or shrapnel in the body),
* patients with tendency toward claustrophobia,
* hemodynamically unstable patients,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-12; Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
blood flow patterns | 2 years
  fluid dynamical properties of blood flow patterns in the heart and surrounding great vessels associated with ethiology of PH

SECONDARY OUTCOMES:
myocardial magnetic relaxation times | 2 years
  left and right ventricular myocardial T1 times associated with ethiology of PH
pulmonary ventilation and perfusion | 2 years
  pulmonary ventilation and perfusion associated with ethiology of PH

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Reiter, PhD, Principal Investigator — Medical Unitersity Graz, Department of Radiology, Division of General Radiology; Michael Fuchsjäger, Prof. Dr., Principal Investigator — Medical Unitersity Graz, Department of Radiology, Division of General Radiology
Locations (1):
- Medical Unitersity Graz, Department of Radiology, Division of General Radiology, Graz, Styria, Austria

REFERENCES:
- [Result] Reiter U, Reiter G, Kovacs G, Stalder AF, Gulsun MA, Greiser A, Olschewski H, Fuchsjager M. Evaluation of elevated mean pulmonary arterial pressure based on magnetic resonance 4D velocity mapping: comparison of visualization techniques. PLoS One. 2013 Dec 12;8(12):e82212. doi: 10.1371/journal.pone.0082212. eCollection 2013. PMID 24349224
- [Result] Reiter G, Reiter U, Kovacs G, Olschewski H, Fuchsjager M. Blood flow vortices along the main pulmonary artery measured with MR imaging for diagnosis of pulmonary hypertension. Radiology. 2015 Apr;275(1):71-9. doi: 10.1148/radiol.14140849. Epub 2014 Nov 5. PMID 25372980
- [Result] Reiter U, Reiter G, Fuchsjager M. MR phase-contrast imaging in pulmonary hypertension. Br J Radiol. 2016 Jul;89(1063):20150995. doi: 10.1259/bjr.20150995. Epub 2016 Apr 6. PMID 26942293
- [Result] Reiter U, Kovacs G, Reiter C, Krauter C, Nizhnikava V, Fuchsjager M, Olschewski H, Reiter G. MR 4D flow-based mean pulmonary arterial pressure tracking in pulmonary hypertension. Eur Radiol. 2021 Apr;31(4):1883-1893. doi: 10.1007/s00330-020-07287-6. Epub 2020 Sep 24. PMID 32974687
- [Result] Reiter G, Kovacs G, Reiter C, Schmidt A, Fuchsjager M, Olschewski H, Reiter U. Left atrial acceleration factor as a magnetic resonance 4D flow measure of mean pulmonary artery wedge pressure in pulmonary hypertension. Front Cardiovasc Med. 2022 Aug 3;9:972142. doi: 10.3389/fcvm.2022.972142. eCollection 2022. PMID 35990987
- [Result] Krauter C, Reiter U, Kovacs G, Reiter C, Masana M, Olschewski H, Fuchsjager M, Stollberger R, Reiter G. Automated vortical blood flow-based estimation of mean pulmonary arterial pressure from 4D flow MRI. Magn Reson Imaging. 2022 May;88:132-141. doi: 10.1016/j.mri.2022.02.007. Epub 2022 Feb 18. PMID 35189283
- [Derived] Reiter G, Reiter U, Kovacs G, Adelsmayr G, Greiser A, Stalder AF, Olschewski H, Fuchsjager M. Counter-clockwise vortical blood flow in the main pulmonary artery in a patient with patent ductus arteriosus with pulmonary arterial hypertension: a cardiac magnetic resonance imaging case report. BMC Med Imaging. 2016 Aug 8;16(1):45. doi: 10.1186/s12880-016-0150-z. PMID 27501792